CLINICAL TRIAL: NCT01445054
Title: A Phase 0 Trial of (111)Indium CHX-A DTPA Trastuzumab Imaging in Cancer
Brief Title: 111 Indium CHX-A DTPA Trastuzumab (Indium-Herceptin) for Imaging Breast Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 070101; 07-C-0101; NCT00474578 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03-07

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer; Colon Cancer
Keywords: 111 Indium Trastuzumab Imaging; PET; Optimal Scanning Strategy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- 1-Arm 1 (Experimental): Subjects with primary or metastatic cancer other than melanoma, basal cell carcinoma, sarcoma, or lymphoma.
  Interventions: Drug: 111Indium CHX-A

INTERVENTIONS:
Drug: 111Indium CHX-A — 111Indium CHX-A will be administered intravenously over a 10-15 minute period using an intravenous catheter

SUMMARY:
Background:

* Some breast cancer cells have specific proteins (receptors) on their surface that make the tumor grow faster than normal cells. One of these receptors is called HER2/neu.
* An FDA-approved drug called Herceptin attaches to HER2/neu if it is present on the cancer cell.
* Indium-Herceptin is an agent in which a tiny amount of radioactivity called Indium has been attached to a tiny amount of Herceptin.

Objectives:

-To see if Indium-Herceptin provides information about the characteristics of the breast cancer in women whose tumors express HER2/neu and those whose tumors do not.

Eligibility:

-Women 18 years or older with primary or metastatic breast cancer who have not received treatment with herceptin for at least 6 months before enrollment into the study.

Design:

* Tissue from the patient s original breast or tumor biopsy is analyzed for HER2/neu status.
* Patients have a physical examination and review of medical records.
* Patients receive an injection of Indium-Herceptin, followed by scanning with a gamma camera that detects the radioactivity in the Indium-Herceptin.
* Patients return to the clinic 1, 2, 3 and 7 days later for repeat imaging to determine the best time to image after injection of Indium-Herceptin.
* Blood samples are obtained every day of scanning to monitor the effects, if any, of the Indium-Herceptin and to see how fast the agent leaves the body.

DETAILED DESCRIPTION:
Background:

* Trastuzumab (Herceptin ), targets HER2 (aka: neu, ErbB2, c-erb-B2) on the surface of cancer cells and is used in the treatment of breast cancers that overexpress HER2/Neu (Erb2). It has also been demonstrated that other malignancies express HER2/Neu (Erb2).
* Radiolabeling trastuzumab could allow human biodistribution studies, noninvasive assessment of HER2/Neu (Erb2) expression, identification of HER2/Neu (Erb2) positive metastases, monitoring of treatment response and establishment of dosimetry for future radioimmunotherapy.
* We have developed a chelated form of trastuzumab, CHX-A DTPA-trastuzumab, that can bind a number of radioisotopes including (111)In, (212), (213)Bi, (212)Pb (86), (90)Y and (177)Lu which have alpha, beta and gamma emissions for imaging and therapy.
* We believe that the agent will be safe based on the low dose of trastuzumab (up to a maximum of 200 mcg of protein or less than1% of the typical loading dose of trastuzumab in a 70 Kg human) and the low dose of radioactivity (5mCi).
* Whereas trastuzumab therapy is generally only useful in tumors that highly express HER2/Neu (Erb2), (111)In-CHX-A DTPA trastuzumab (henceforth (111)Indium-trastuzumab ) will image tumors that are not only highly expressing HER2/Neu (Erb2) but also tumors that are poorly expressing HER2/Neu (Erb2) as documented by preclinical data.

Objectives:

-The primary objective is to compare uptake of 111Indium trastuzumab with HER2/Neu (Erb2) status of the tumor as determined by IHC

Eligibility:

* Participants with a history of primary or metastatic cancer (other than melanoma, basal cell carcinoma, sarcoma or lymphoma) with known solid tumor size greater than or equal to 1.5 cm.
* Availability of HER2/Neu (Erb2) expression by immunohistochemistry (IHC) or pathology or biopsy specimen can be provided on which such an analysis can be made.

Design:

* The design of this pilot trial follows the concept of a Phase 0 or Exploratory IND (xIND) study.
* Participants with known malignancy greater than or equal to 1.5cm and known HER2/Neu(ErbB2) tumor status (0, 1+, 2+ or 3+) by IHC or FISH.
* After receiving 5 mCi of (111)Indium-trastuzumab, all participants will undergo gamma camera scans at approximately 24-72 hours after injection. In some subjects, an additional imaging session may be required 24 hours after the first set of images as physiologic bowel clearance is variable and may obscure the lesion of interest on the initial scan.
* We will accrue 20 participants to this study.
* A total of 8 blood samples (4 lab tests and up to 4 for pharmacokinetics) will be obtained from each participant to establish toxicity and the pharmacokinetics of clearance.
* Images will be correlated with IHC status using tumor to background ratios and the optimal scanning strategy with regard to HER2/neu(ErbB2) expression will be determined.
* Participants who undergo a therapy thought to target or effect HER2 will have the option of undergoing repeat imaging following therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participant must have histological confirmation of primary or metastatic cancer other than melanoma, basal cell carcinoma, sarcoma, or lymphoma.

* Primary tumor or metastatic focus must be 1.5cm or greater in diameter as established by palpation, ultrasound, mammography, CT or MRI.
* Participant must be 18 years or older.
* Availability of tumor tissue (either from the initial primary tumor or from current tumor lesion) for performing IHC or FISH analysis for HER2/Neu (Erb2)
* Chemistry and CBC parameters: serum creatinine less than or equal to 1.4mg/dl. SGOT and SGPT less than or equal to 3 times of the upper limits of normal; total bilirubin, of less than or equal to 2 times the upper limits of normal or 3.0 mg/dl in patients with Gilbert s syndrome; platelet count must be greater than 100,00.
* ECOG Performance score of 0 or 1.
* Ability to provide informed consent.
* Negative serum pregnancy test (within 48 hours of imaging agent injection) in women of child bearing age and willingness to use contraception (barrier, abstinence, non-hormonal) for 3 weeks after injection of (111)Indium trastuzumab if participant is of child bearing age.

EXCLUSION CRITERIA:

* Known allergy to trastuzumab.
* Pregnant or lactating women.
* Participants for whom enrollment would significantly delay (greater than 2 weeks) the scheduled standard of care therapy.
* Participants with an active second malignancy (excluding treated basal cell skin carcinoma).
* History of cardiac disease (myocardial infarction, arrhythmias requiring therapy, symptomatic valvular disease, cardiomyopathy, or pericarditis).
* Participants with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Participants with severe claustrophobia.
* A participant who needs a nuclear medicine scan other than a PET scan as part of their work-up cannot enroll until these scans have been completed.
* Gamma-camera table restrictions preclude scanning participants greater than 350 lbs (160 Kg)
* With the exception of AT13387 and PU-H71, and Ad5f35HER2ECTM transduced autologous dendritic cell vaccine participants cannot have received another experimental drug within 14 days prior to or during study enrollment.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-03-01; Primary Completion 2014-08-20 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
Compare uptake of 111Indium-CHX-A DTPA trastuzumab with HER2/Neu (ErbB2) status of the tumor as determined by IHC | 5 days after intervention
  Correlation between uptake of 111Indium-CHX-A DTPA trastuzumab with HER2/Neu (ErbB2) and status of the tumor as determined by IHC

SECONDARY OUTCOMES:
Safety of 111Indium-trastuzumab. | 30 days after intervention
  List of adverse event frequency
Optimal timing of 111Indium-CHX-A DTPA trastuzumab imaging as a function of HER2/ Neu(ErbB2) status. | completion of study
  Optimal timing of 111Indium-CHX-A DTPA trastuzumab imaging as a function of HER2/ Neu(ErbB2) status.
Biodistribution of the agent in normal organs | completion of study
  Biodistribution of the agent in normal organs
Pharmacokinetic serum clearance of 111Indium-CHXA DTPA trastuzumab | 24 hours after intervention
  Drug level in blood
To evaluate the change in 111Indium-CHX-A DTPA trastuzumab uptake in tumors following treatment with a HER2 targeted therapy | completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Choyke, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Milenic DE, Garmestani K, Brady ED, Albert PS, Ma D, Abdulla A, Brechbiel MW. Targeting of HER2 antigen for the treatment of disseminated peritoneal disease. Clin Cancer Res. 2004 Dec 1;10(23):7834-41. doi: 10.1158/1078-0432.CCR-04-1226. PMID 15585615
- [Background] Pegram MD, Pauletti G, Slamon DJ. HER-2/neu as a predictive marker of response to breast cancer therapy. Breast Cancer Res Treat. 1998;52(1-3):65-77. doi: 10.1023/a:1006111117877. PMID 10066073
- [Background] Menard S, Casalini P, Campiglio M, Pupa S, Agresti R, Tagliabue E. HER2 overexpression in various tumor types, focussing on its relationship to the development of invasive breast cancer. Ann Oncol. 2001;12 Suppl 1:S15-9. doi: 10.1093/annonc/12.suppl_1.s15. PMID 11521715